CLINICAL TRIAL: NCT07085962
Title: A Randomized, Controlled Study to Evaluate the Efficacy and Safety of Calculus Bovis Sativus in Adult Subjects With Metabolic Dysfunction-associated Fatty Liver Disease (MAFLD)
Brief Title: Efficacy and Safety of Calculus Bovis Sativus in Adults With MAFLD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Cheng, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBS-MAFLD-2025
Record Dates: First submitted 2025-06-12; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Dysfunction-associated Fatty Liver Disease
Keywords: metabolic dysfunction-associated fatty liver disease; Calculus bovis sativus; Hypertransaminasemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calculus bovis sativus group (Experimental): Participants will receive Calculus bovis sativus 200mg orally, once daily (qd) for 12 weeks.
  Interventions: Drug: Calculus bovis sativus
- placebo group (Placebo Comparator): Participants will receive placebo matched in appearance, taste, and smell to the active drug, orally, once daily (qd) for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calculus bovis sativus — Calculus bovis sativus 200mg qd
  Arms: Calculus bovis sativus group
Drug: Placebo — Placebo 200mg qd
  Arms: placebo group

SUMMARY:
Metabolic dysfunction-associated fatty liver disease (MAFLD) has become the most common chronic liver disease worldwide. Timely therapeutic intervention for MAFLD is crucial for improving patient prognosis and preventing its progression to liver fibrosis, cirrhosis, and even hepatocellular carcinoma (HCC). Therefore, the discovery of novel drugs for the treatment of MAFLD is of great significance.

Previous clinical studies have shown that calculus bovis sativus, as an adjuvant therapy for icteric hepatitis and chronic hepatitis B, exhibits significant anti-inflammatory and enzyme-reducing effects, improves liver function indicators, and enhances overall clinical outcomes. However, there is currently no clinical research on the therapeutic effects of calculus bovis sativus in patients with MAFLD, and its underlying mechanisms of action remain to be elucidated.

This study proposes a randomized, double-blind, placebo-controlled trial to investigate the effects of calculus bovis sativus in adult patients with MAFLD. The primary objective is to preliminarily explore the clinical efficacy of calculus bovis sativus in treating MAFLD, particularly its impact on liver injury and inflammation. Furthermore, this research will employ a multi-omics approach, integrating metagenomics and metabolomics, to analyze the effects of calculus bovis sativus on the gut microbiota and their metabolites in MAFLD patients. The aim is to uncover its potential mechanisms of action, thereby facilitating its clinical translation and application, and ultimately providing a new therapeutic strategy for patients with MAFLD.

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, placebo-controlled trial to investigate calculus bovis sativus in adult subjects with metabolic dysfunction-associated fatty liver disease (MAFLD). The study aims to evaluate the safety of calculus bovis sativus in subjects with MAFLD by monitoring the incidence of adverse events and key laboratory parameters, including routine blood and urine tests, as well as hepatic and renal function, and to preliminarily investigate the potential clinical efficacy of calculus bovis sativus in mitigating MAFLD, liver injury, and inflammation by monitoring various serum biomarkers and non-invasive assessment parameters, such as the controlled attenuation parameter (CAP), liver stiffness measurement (LSM), and magnetic resonance imaging proton density fat fraction (MRI-PDFF). Furthermore, this study will employ a multi-omics approach, combining metagenomics and metabolomics, to explore the effects of calculus bovis sativus on the gut microbiota and its metabolites in patients with MAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the informed consent form (ICF) prior to the study and is fully aware of the study's content, procedures, and potential adverse reactions.
2. Is able to complete the study in accordance with the protocol requirements.
3. The subject (and/or partner) agrees to use effective contraceptive measures voluntarily from the screening period until 6 months after the last dose of the investigational product.
4. At the time of signing the ICF, age is between 18 and 75 years (inclusive), with no restriction on sex.
5. Meets the diagnostic criteria outlined in the "Guidelines for the Prevention and Treatment of Metabolic Dysfunction-Associated (Non-alcoholic) Fatty Liver Disease (2024 Edition)" issued by the Chinese Society of Hepatology, Chinese Medical Association.
6. Confirmed significant hepatic steatosis by transient elastography (Fibroscan) with a Controlled Attenuation Parameter (CAP) value ≥ 240 dB/m.
7. Liver enzyme levels meet the following criteria: 1 × upper limit of normal (ULN) < serum AST and ALT < 5 × ULN.
8. Exclusion of significant liver fibrosis based on non-invasive assessment, meeting at least one of the following four conditions:

   * FIB-4 < 1.3
   * NAFLD Fibrosis Score (NFS) < -1.455
   * LSM < 8.0 kPa
   * FAST score < 0.35
9. Stable body weight for at least 6 weeks prior to screening, defined as a weight change (increase or decrease) of ≤5%.

Exclusion Criteria:

1. Presence of the following chronic diseases: viral hepatitis; positive serology for Human Immunodeficiency Virus (HIV); primary sclerosing cholangitis, primary biliary cholangitis, autoimmune hepatitis, drug-induced liver disease, alcoholic liver disease, or Wilson's disease.
2. Excessive alcohol consumption (defined as >30g of alcohol per day for males or >20g per day for females).
3. History of diabetes other than type 2 diabetes, such as type 1 diabetes, secondary diabetes, etc.
4. History of malignancy (except for those with a tumor-free period of more than 5 years prior to screening), or currently under evaluation for active or suspected malignancy. Exceptions include fully treated basal cell carcinoma, squamous cell skin carcinoma, or cervical carcinoma in situ.
5. History of bariatric surgery within the 5 years prior to screening (inclusive).
6. Use of antibiotics within the last 3 weeks or during the study period.
7. Underwent major surgery within 3 months prior to signing the ICF, or planning to undergo major surgery during the study period. (Major surgery is defined as a procedure with risk to the patient's life, particularly surgery involving the cranium, chest, abdomen, or pelvic organs).
8. Recent history of drug abuse (defined as ≤2 years).
9. Presence of psychosis or any other cognitive impairment, or other conditions that would interfere with the subject's compliance.
10. Currently receiving any approved therapy for MASH. Receiving anticoagulant therapy (e.g., warfarin, heparin), or participated in another interventional clinical trial with a drug product within 3 months prior to screening.
11. Presence of any of the following laboratory exclusion criteria at screening (the study center may repeat the test once for any abnormal value):

    * Serum ALT or AST > 5 × ULN
    * Alkaline phosphatase (ALP) ≥ 2 × ULN
    * eGFR < 60 mL/min
    * Total bilirubin > 1.5 × ULN
    * Platelet count < lower limit of normal (LLN)
12. Received a blood transfusion within ≤2 months prior to screening and/or donated blood within ≤1 month prior to screening. Note: Subjects are not permitted to donate blood throughout the entire study period.
13. Presence of portal hypertension, such as esophageal varices, ascites, or hepatic encephalopathy.
14. Pregnant or lactating females.
15. History of liver transplantation or planned liver transplantation.
16. Presence of any significant systemic or major diseases other than liver disease, including recent (≤6 months prior to screening) congestive heart failure (New York Heart Association [NYHA] Functional Classification III-IV), unstable coronary artery disease, arterial revascularization, respiratory disease, renal failure, stroke, transient ischemic attack, organ transplant, psychiatric disorders, or any other clinically significant disease-related event requiring hospitalization within 6 months prior to screening.
17. Acute or chronic gastrointestinal diseases (including diarrhea, gastrointestinal infections, inflammatory bowel disease, etc.).
18. Any condition that, in the opinion of the investigator, would pose a safety risk to the subject or may interfere with the conduct of the study, or if the investigator believes the subject is unlikely to complete the study or comply with its requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Alanine Aminotransferase (ALT) at Week 12 | At baseline and after 4 weeks,8 weeks and 12 weeks of treatment
  Alanine Aminotransferase (ALT) will be measured from serum samples. The result will be reported in international units per liter (U/L).

SECONDARY OUTCOMES:
Change from Baseline in Aspartate Aminotransferase (AST) at Week 12 | Baseline, Week 4, Week 8, and Week 12
  Aspartate Aminotransferase (AST) will be measured from serum samples. The result will be reported in international units per liter (U/L).
Change from Baseline in Gamma-glutamyl Transferase (GGT) at Week 12 | At baseline and after 4 weeks,8 weeks and 12 weeks of treatment
  Gamma-glutamyl Transferase (GGT) will be measured from serum samples. The result will be reported in international units per liter (U/L).
Change from Baseline in Total Bilirubin at Week 12 | At baseline and after 4 weeks,8 weeks and 12 weeks of treatment
  Total Bilirubin will be measured from serum samples. The result will be reported in micromoles per liter (μmol/L).
Change from Baseline in Alkaline Phosphatase (ALP) at Week 12 | At baseline and after 4 weeks,8 weeks and 12 weeks of treatment
  Alkaline Phosphatase (ALP) will be measured from serum samples. The result will be reported in international units per liter (U/L).
Change from Baseline in Liver Stiffness Measurement (LSM) by Fibroscan at Week 12 | At baseline and after 12 weeks of treatment
  Liver Stiffness Measurement (LSM) is assessed using Fibroscan to evaluate liver fibrosis. The result is reported in kilopascals (kPa).
Change from Baseline in Controlled Attenuation Parameter (CAP) by Fibroscan at Week 12 | At baseline and after 12 weeks of treatment
  Controlled Attenuation Parameter (CAP) is assessed using Fibroscan to quantify liver steatosis (fat content). The result is reported in decibels per meter (dB/m).
Change from Baseline in Body Weight at Week 12 | At baseline and after 12 weeks of treatment
  Body weight will be measured in kilograms (kg).
Change from Baseline in Body Mass Index (BMI) at Week 12 | At baseline and after 12 weeks of treatment
  Body Mass Index (BMI) is calculated as weight in kilograms divided by the square of height in meters (kg/m²).
Change from Baseline in Waist Circumference at Week 12 | At baseline and after 12 weeks of treatment
  Waist circumference will be measured in centimeters (cm).
Change from Baseline in Hip Circumference at Week 12 | At baseline and after 12 weeks of treatment
  Hip circumference will be measured in centimeters (cm)
Change from Baseline in Fasting Blood Glucose (FBG) at Week 12 | At baseline and after 12 weeks of treatment
  Fasting Blood Glucose (FBG) will be measured from plasma samples. The result will be reported in millimoles per liter (mmol/L).
Change from Baseline in Glycated Hemoglobin (HbA1c) at Week 12 | At baseline and after 12 weeks of treatment
  Glycated Hemoglobin (HbA1c) will be measured from whole blood samples. The result will be reported as a percentage (%)
Change from Baseline in Fasting Insulin at Week 12 | At baseline and after 12 weeks of treatment
  Fasting insulin will be measured from serum samples. The result will be reported in micro-international units per milliliter (μIU/mL).
Change from Baseline in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) at Week 12 | At baseline and after 12 weeks of treatment
  The Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) is a calculated index based on fasting glucose and fasting insulin. It is calculated using the formula: [Fasting Insulin (μIU/mL) x Fasting Glucose (mmol/L)] / 22.5.
Change from Baseline in Total Cholesterol (TC) at Week 12 | At baseline and after 12 weeks of treatment
  Total Cholesterol (TC) will be measured from serum samples. The result will be reported in millimoles per liter (mmol/L).
Change from Baseline in Triglycerides (TG) at Week 12 | At baseline and after 12 weeks of treatment
  Triglycerides (TG) will be measured from serum samples. The result will be reported in millimoles per liter (mmol/L).
Change from Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at Week 12 | At baseline and after 12 weeks of treatment
  High-Density Lipoprotein Cholesterol (HDL-C) will be measured from serum samples. The result will be reported in millimoles per liter (mmol/L).
Change from Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12 | At baseline and after 12 weeks of treatment
  Low-Density Lipoprotein Cholesterol (LDL-C) will be measured from serum samples. The result will be reported in millimoles per liter (mmol/L).
Change from Baseline in Liver Fat Fraction as Measured by MRI-PDFF at Week 12 | At baseline and after 12 weeks of treatment
  Liver fat fraction will be quantified using Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF)
Change from Baseline in Gut Microbiota Alpha Diversity as Measured by the Shannon Index at Week 12 | At baseline and after 12 weeks of treatment
  Gut microbiota composition will be analyzed from stool samples using 16S rRNA sequencing. Alpha diversity, a measure of within-sample microbial richness and evenness, will be calculated using the Shannon index.
Change from Baseline in Fecal Short-Chain Fatty Acid (SCFA) Concentrations at Week 12 | At baseline and after 12 weeks of treatment
  Concentrations of key Short-Chain Fatty Acids (SCFAs), such as butyrate and propionate, will be quantified from stool samples using mass spectrometry-based metabolomics.
Change from Baseline in Serum Total Bile Acid (TBA) Concentration at Week 12 | At baseline and after 12 weeks of treatment
  Serum Total Bile Acid (TBA) concentration will be quantified using mass spectrometry-based metabolomics.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) as Graded by CTCAE v6.0 | From Baseline up to Week 12
  A Treatment-Emergent Adverse Event (TEAE) is defined as any adverse event occurring or worsening on or after the first dose of the study drug up to the final study visit at Week 12. The severity of all TEAEs will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) v6.0.
Change from Baseline in Platelet Count at Week 12 | At baseline and after 4 weeks,8 weeks and 12 weeks of treatment
  Platelet count will be measured from a whole blood sample as part of routine safety monitoring. The result will be reported in gigaparticles per liter (x10^9/L).
Change from Baseline in Serum Creatinine at Week 12 | At baseline and after 4 weeks,8 weeks and 12 weeks of treatment
  Serum creatinine will be measured from a blood sample as part of routine safety monitoring. The result will be reported in micromoles per liter (μmol/L).
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 12 | At baseline and after 4 weeks,8 weeks and 12 weeks of treatment
  The Estimated Glomerular Filtration Rate (eGFR) is calculated based on serum creatinine, age, and sex, using the CKD-EPI 2021 equation. It is a key indicator of kidney function, reported in mL/min/1.73 m².

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cheng, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No